CLINICAL TRIAL: NCT03673306
Title: A Multicenter Retrospective Study on the Prognostic Impact of Pregnancy in Women With History of BRCA Mutated Breast Cancer
Brief Title: Safety of Pregnancy in BRCA Mutated Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IJB-BRCAPreg-CE2630
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; BRCA; Young; Survivorship
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant cohort: Women with one or more pregnancies any time after breast cancer diagnosis
  Interventions: Other: Clinical outcomes
- Non-pregnant cohort: Women with no subsequent pregnancies after breast cancer diagnosis
  Interventions: Other: Clinical outcomes

INTERVENTIONS:
Other: Clinical outcomes — Clinical outcomes

SUMMARY:
The present study aims at refining the understanding of the effect of pregnancy on breast cancer outcomes in the specific population of BRCA mutated patients with known history of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive breast cancer between January 2000 and December 2020;
* Breast cancer diagnosis at the age of ≤ 40 years;
* Known presence of germline BRCA mutation.

Exclusion Criteria:

* Known BRCA mutation with no diagnosis of invasive breast cancer;
* Diagnosis of ovarian cancer or other malignancies with no history of invasive breast cancer;
* Diagnosis of hereditary or familiar invasive breast cancer without BRCA mutation or with BRCA genes not tested;
* Diagnosis of invasive breast cancer with germline BRCA variants of unknown significance.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women only
Study Population: Patients with diagnosis of invasive breast cancer between January 2000 and December 2020 at the age of ≤ 40 years and with known presence of germline BRCA mutation.
Sampling Method: Probability Sample
Enrollment: 4732 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (81):
- United States (7):
  - Yale University, New Haven, Connecticut
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Michigan State University, Lansing, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Lifespan Cancer Institute, Providence, Rhode Island
- Argentina (3):
  - Hospital Aleman, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
- Australia (2):
  - kConFab, Follow-up Project, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Medical University of Vienna, Vienna, Austria
- Belgium (3):
  - Cliniques Universitaires Saint-Luc UCL, Brussels
  - Institut Jules Bordet, Brussels
  - University Hospitals Leuven, KU Leuven, Leuven
- Clinical Center University of Sarajevo, Sarajevo, Bosnia and Herzegovina
- Brazil (2):
  - Hospital Sírio-Libanês, Brasília
  - Cancer Institute ICESP, São Paulo
- Mc Gill University, Montreal, Canada
- France (6):
  - Bergonie Institute, Bordeaux
  - Leon Berard Cancer Center, Lyon
  - Hopital Saint Louis, Paris
  - Institut Curie, Paris
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif
- Todua Clinic, Tbilisi, Georgia
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Leitung, Brustzentrum der Universität München (LMU), München
- Tata Memorial Centre, Mumbai, India
- Israel (4):
  - Sharett Institute of Oncology - Hadassah Hebrew University Medical Center, Jerusalem
  - Davidoff Cancer Center - Rabin Medical Center - Beilinson, Petah Tikva
  - Sheba Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (22):
  - Università Politecnica delle Marche - Azienda Ospedaliero-Universitaria Ospedali Riuniti Umberto I - GM Lancisi - G Salesi, Ancona
  - Oncological Center CRO, Aviano
  - Azienda Ospedaliera "Papa Giovanni XXIII", Bergamo
  - Azienda Ospedaliero Universitaria di Cagliari, Cagliari
  - Candiolo Cancer Center (IRCCS), Candiolo
  - Florence University Hospital - University of Florence, Florence
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Azienda USL Toscana Sud Est - Misericordia Hospital, Grosseto
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori (IRST) Dino Amadori, Meldola
  - European Institute of Oncology, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria Policlinico, University of Modena and Reggio Emilia, Modena
  - San Gerardo Hospital ASST Monza, Monza
  - University of Naples "Federico II", Naples
  - IOV (Istituto Oncologico Veneto), Padua
  - IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana - Ospedale Santa Chiara, Pisa
  - Nuovo Ospedale di Prato - Santo Stefano, Prato
  - AOU Policlinico Umberto I, Roma
  - ASL Roma 1 - Centro Oncologico S. Spirito - Nuovo Regina Margherita, Rome
  - Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Saint Joseph University of Beirut, Beirut, Lebanon
- Mexico (2):
  - Instituto Nacional de Cancerologia, Mexico City
  - Hospital Zambrano Hellion - Tecnologico de Monterrey, Monterrey
- Netherlands Cancer Institute, Amsterdam, Netherlands
- Poland (4):
  - Medical University of Gdansk, Gdansk
  - Poznan University of Medical Sciences, University Hospital of H. Swiecicki, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
  - Military institute of Medicine, Warsaw
- Portugal (2):
  - Champalimaud Foundation, Lisbon
  - Hospital de Santa Maria and Instituto de Medicina Molecular of the Faculty of Medicine of the University of Lisbon, Lisbon
- Institute of Oncology "Ion Chiricuta", Cluj-Napoca, Romania
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Oncology Institute of Vojvodina - University of Novi Sad, Novi Sad
- St. Elisabeth Cancer Institute (Onkologicky ustav sv. Alzbety-OUSA), Bratislava, Slovakia
- University of Ulsan, College of Medicine, Asan medical center, Seoul, South Korea
- Spain (6):
  - Hospital Clínic of Barcelona, Barcelona
  - Vall D'Hebron University Hospital, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Ramon y Cajal - IOB Institute of Oncology (Madrid) - International Breast Cancer Center (IBCC), Madrid
  - Hospital Universitari Son Espases Palma, Palma de Mallorca
  - INCLIVA, University Hospital of Valencia, Valencia
- Sweden (3):
  - Capio Saint Göran's Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Stockholm Southern Hospital (Södersjukhuset), Stockholm
- Oncology Institute of Southern Switzerland, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Result] Lambertini M, Ameye L, Hamy AS, Zingarello A, Poorvu PD, Carrasco E, Grinshpun A, Han S, Rousset-Jablonski C, Ferrari A, Paluch-Shimon S, Cortesi L, Senechal C, Miolo G, Pogoda K, Perez-Fidalgo JA, De Marchis L, Ponzone R, Livraghi L, Estevez-Diz MDP, Villarreal-Garza C, Dieci MV, Clatot F, Berliere M, Graffeo R, Teixeira L, Cordoba O, Sonnenblick A, Luna Pais H, Ignatiadis M, Paesmans M, Partridge AH, Caron O, Saule C, Del Mastro L, Peccatori FA, Azim HA Jr. Pregnancy After Breast Cancer in Patients With Germline BRCA Mutations. J Clin Oncol. 2020 Sep 10;38(26):3012-3023. doi: 10.1200/JCO.19.02399. Epub 2020 Jul 16. PMID 32673153
- [Result] Lambertini M, Blondeaux E, Agostinetto E, Hamy AS, Kim HJ, Di Meglio A, Bernstein Molho R, Hilbers F, Pogoda K, Carrasco E, Punie K, Bajpai J, Ignatiadis M, Moore HCF, Phillips KA, Toss A, Rousset-Jablonski C, Peccatori FA, Renaud T, Ferrari A, Paluch-Shimon S, Fruscio R, Cui W, Wong SM, Vernieri C, Ruddy KJ, Dieci MV, Matikas A, Rozenblit M, Villarreal-Garza C, De Marchis L, Del Mastro L, Puglisi F, Del Pilar Estevez-Diz M, Rodriguez-Wallberg KA, Mrinakova B, Meister S, Livraghi L, Clatot F, Yerushalmi R, De Angelis C, Sanchez-Bayona R, Meattini I, Cichowska-Cwalinska N, Berliere M, Salama M, De Giorgi U, Sonnenblick A, Chiodi C, Lee YJ, Maria C, Azim HA Jr, Boni L, Partridge AH; BRCA BCY Collaboration. Pregnancy After Breast Cancer in Young BRCA Carriers: An International Hospital-Based Cohort Study. JAMA. 2024 Jan 2;331(1):49-59. doi: 10.1001/jama.2023.25463. PMID 38059899
- [Derived] Blondeaux E, Sonnenblick A, Agostinetto E, Bas R, Kim HJ, Franzoi MA, Bernstein-Molho R, Linn S, Kwong A, Pogoda K, Balmana J, Smeets A, Bajpai J, Moore HCF, Partridge AH, Phillips KA, Toss A, Rousset-Jablonski C, Peccatori FA, Renaud T, Ferrari A, Paluch-Shimon S, Mando P, Lee JE, Fruscio R, Cui W, Wong SM, Vernieri C, Ruddy KJ, Dieci MV, Matikas A, Rozenblit M, Guven DC, Lee M, Villarreal-Garza C, Hwang SE, De Marchis L, Puglisi F, Kemp Z, Meireles PA, Parokonnaya A, Werutsky G, Okano M, Azim HA Jr, Mati K, Rosenberg S, Gelber R, Boni L, Lambertini M. Association between risk-reducing surgeries and survival in young BRCA carriers with breast cancer: an international cohort study. Lancet Oncol. 2025 Jun;26(6):759-770. doi: 10.1016/S1470-2045(25)00152-4. Epub 2025 May 8. PMID 40347973
- [Derived] Lambertini M, Blondeaux E, Tomasello LM, Agostinetto E, Hamy AS, Kim HJ, Franzoi MA, Bernstein-Molho R, Hilbers F, Pogoda K, Wildiers H, Bajpai J, Ignatiadis M, Moore HCF, Partridge AH, Phillips KA, Toss A, Rousset-Jablonski C, Criscitiello C, Renaud T, Ferrari A, Paluch-Shimon S, Fruscio R, Cui W, Wong SM, Vernieri C, Ruddy KJ, Dieci MV, Matikas A, Rozenblit M, Villarreal-Garza C, De Marchis L, Puglisi F, Rodriguez-Wallberg KA, Duhoux FP, Livraghi L, Bruzzone M, Boni L, Balmana J. Clinical Behavior of Breast Cancer in Young BRCA Carriers and Prediagnostic Awareness of Germline BRCA Status. J Clin Oncol. 2025 May 10;43(14):1706-1719. doi: 10.1200/JCO-24-01334. Epub 2025 Feb 24. PMID 39993249
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32673153/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/38059899/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects should meet all eligibility criteria and have available information on pregnancy status before assignment to groups
Period: Overall Study
Arm/Group | Pregnant Cohort | Non-pregnant Cohort
Started | 659 | 4073
Completed | 659 | 4073
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnant Cohort | Non-pregnant Cohort | Total
Number analyzed (Participants) | 659 | 4073 | 4732
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [28 to 33] | 35 [32 to 38] | 35 [31 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 659 | 4073 | 4732
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: The primary end points were the cumulative incidence of pregnancy and disease-free survival.
Time Frame: 10 years
Population: A disease-free survival event was defined as the occurrence of 1 of the following invasive events: locoregional recurrence, distant metastases, new contralateral or ipsilateral invasive breast cancer, second primary malignancy, or death due to any cause.
Measure: Number; unit: DFS events/100*person-year
Arm/Group | Pregnant Cohort | Non-pregnant Cohort
Number analyzed (Participants) | 659 | 4073
DFS events/100*person-year | 5.44 | 5.45

2. Primary Outcome: Cumulative Incidence of Pregnancy After Breast Cancer
Description: The primary end points were the cumulative incidence of pregnancy and disease-free survival.
Time Frame: 10 years
Measure: Number (95% Confidence Interval); unit: Percentage (Cumulative incidence at 10y)
Groups:
- Overall Cohort: Overall cohort
Arm/Group | Overall Cohort
Number analyzed (Participants) | 4732
Percentage (Cumulative incidence at 10y) | 22 [21 to 24]

3. Secondary Outcome: Breast Cancer-Specific Survival
Description: A breast cancer-specific survival event was defined as death due to breast cancer, and patients who died for reasons other than breast cancer were censored at the date of death.
Time Frame: 10 years
Population: Breast cancer-specific survival
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Cohort | Non-pregnant Cohort
Number analyzed (Participants) | 659 | 4073
Participants | 35 | 523

4. Secondary Outcome: Overall Survival
Description: An overall survival event was defined as death due to any cause.
Time Frame: 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Cohort | Non-pregnant Cohort
Number analyzed (Participants) | 659 | 4073
Participants | 39 | 570

ADVERSE EVENTS:
Time Frame: 10 years
Description: All-Cause Mortality was recorded and is reported below. Adverse events were not collected. Please consider that this is a restrospective, observational study. No intervention was performed.
Groups:
- Pregnancy Cohort: Women with one or more pregnancies any time after breast cancer diagnosis
- No Pregnancy Cohort: Women with no pregnancies after breast cancer diagnosis
Arm/Group | Pregnancy Cohort | No Pregnancy Cohort
All-Cause Mortality (participants affected / at risk) | 39/659 | 570/4073
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03673306/Prot_SAP_000.pdf